CLINICAL TRIAL: NCT06237114
Title: Phase II Clinical Trial to Evaluate the Early Return of Urinary Continence Utilizing a Novel Hybrid Transvesical Adapted Retzius Sparing Robotic Assisted Radical Prostatectomy Technique
Brief Title: Novel Robotic Prostatectomy Technique for Early Urinary Continence
Acronym: TRS-RALP
Status: Completed | Type: Observational
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Victor McPherson, MD, MSc, FRCSC, Assistant Professor Division of Urology, Sir Mortimer B. Davis - Jewish General Hospital
Other Study IDs: 2024-3985
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this a single arm prospective study is to evaluating the 3-month return of urinary continence outcomes of patients undergoing the transvesical retzius sparing robotic radical prostatectomy (TRS-RALP) for standard of care surgical prostate removal for treatment of prostate cancer.

The main question it aims: To have patients respond to questionnaires to collect exploratory data on patient's quality of life (QoL; EuroQol-5 Dimension 5-Level [EQ-5D-5L] and prostate cancer related urinary, bowel, and sexual function questionnaires (Expanded Prostate cancer Index Composite for Clinical Practice (EPIC-CP), at their standard of care perioperative visits at baseline and at 4 weeks, 3- and 6-months post operatively.

DETAILED DESCRIPTION:
Patients undergoing robotic prostatectomy will have their surgery performed utilizing TRS-RALP technique, which is a novel combination of two previously described techniques. This technique is a recent alteration to our standard of care method of prostate removal, and comprises two halves of two previously validated techniques performed in succession. No new safety signals are anticipated, and the technique has been in use since May 2023. The purpose of this technique change is to improve the rate of return urinary continence, which early institutional experience supports. This trial protocol has been generated to formally evaluate this continence return improvement inside a statistical framework for prospective verification in our entire patient cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing standard of care robotic radical prostatectomy for localized prostate cancer

Exclusion Criteria:

* Patients with previous pelvic surgery
* Patients with previous pelvic radiotherapy
* Patient with previous focal therapy for prostate cancer
* Patients aged < 18 years at diagnosis
* Legally incapable patients
* Patients who are unable to receive information about the study in a language they understand
* Patients who are unable to complete questionnaires and have no companion to help complete them
* Patients undergoing a concomitant cancer surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Study Population: Urology clinic at the the hospital
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-03-08 (Actual); Primary Completion 2025-03-08 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
EQ-5D-5L #1.1 | Pperioperative baseline
  The EuroQol - 5 Dimension - 5 Level is a questionnaire that provides a descriptive profile for health status. The questionnaire is comprised of 5 dimension questions; mobility, self care, usual activities, pain/discomfort, anxiety/depression. For each dimension, the patient is asked to check off a level associated; no problems, slight problems, moderate problems, severe problems, extreme problems. Each result is a 1-digit number expressing the level of that dimension. The final result is a 5 digit number describing the patient's health state. The digits range from 1 (best health - best possible outcome) to 5 (worst health - worst possible outcome).
  The final question asks the patient to check their current health status. This ranges from 100 (best health you can imagine - best outcome) to 0 (worst health you can imagine - worst outcome).
EQ-5D-5L #1.2 | 4 weeks postoperatively
  The EuroQol - 5 Dimension - 5 Level is a questionnaire that provides a descriptive profile for health status. The questionnaire is comprised of 5 dimension questions; mobility, self care, usual activities, pain/discomfort, anxiety/depression. For each dimension, the patient is asked to check off a level associated; no problems, slight problems, moderate problems, severe problems, extreme problems. Each result is a 1-digit number expressing the level of that dimension. The final result is a 5 digit number describing the patient's health state. The digits range from 1 (best health - best possible outcome) to 5 (worst health - worst possible outcome).
  The final question asks the patient to check their current health status. This ranges from 100 (best health you can imagine - best outcome) to 0 (worst health you can imagine - worst outcome).
EQ-5D-5L #1.3 | 3 months postoperatively
  The EuroQol - 5 Dimension - 5 Level is a questionnaire that provides a descriptive profile for health status. The questionnaire is comprised of 5 dimension questions; mobility, self care, usual activities, pain/discomfort, anxiety/depression. For each dimension, the patient is asked to check off a level associated; no problems, slight problems, moderate problems, severe problems, extreme problems. Each result is a 1-digit number expressing the level of that dimension. The final result is a 5 digit number describing the patient's health state. The digits range from 1 (best health - best possible outcome) to 5 (worst health - worst possible outcome).
  The final question asks the patient to check their current health status. This ranges from 100 (best health you can imagine - best outcome) to 0 (worst health you can imagine - worst outcome).
EQ-5D-5L #1.4 | 6 months postoperatively
  The EuroQol - 5 Dimension - 5 Level is a questionnaire that provides a descriptive profile for health status. The questionnaire is comprised of 5 dimension questions; mobility, self care, usual activities, pain/discomfort, anxiety/depression. For each dimension, the patient is asked to check off a level associated; no problems, slight problems, moderate problems, severe problems, extreme problems. Each result is a 1-digit number expressing the level of that dimension. The final result is a 5 digit number describing the patient's health state. The digits range from 1 (best health - best possible outcome) to 5 (worst health - worst possible outcome).
  The final question asks the patient to check their current health status. This ranges from 100 (best health you can imagine - best outcome) to 0 (worst health you can imagine - worst outcome).
EPIC-CP #2.1 | perioperative baseline
  The Expanded Prostate cancer Index Composite for Clinical Practice is a questionnaire to measure urinary, bowel,sexual and hormonal function of the patient's prostate cancer quality of life. The questionnaire is scored by the sum of the following scores: Urinary Incontinence symptom score, Urinary Irritation/Obstructive symptom score, Bowel Symptom score, Vitality/Hormonal symptom score and the overall prostate cancer quality of life score. The range of the score varies from 0 (best possible outcome) to 60 (worst possible outcome).
Expanded Prostate cancer Index Composite for Clinical Practice (EPIC-CP) #2.2 | 4 weeks postoperatively
  The Expanded Prostate cancer Index Composite for Clinical Practice is a questionnaire to measure urinary, bowel,sexual and hormonal function of the patient's prostate cancer quality of life. The questionnaire is scored by the sum of the following scores: Urinary Incontinence symptom score, Urinary Irritation/Obstructive symptom score, Bowel Symptom score, Vitality/Hormonal symptom score and the overall prostate cancer quality of life score. The range of the score varies from 0 (best possible outcome) to 60 (worst possible outcome).
Expanded Prostate cancer Index Composite for Clinical Practice (EPIC-CP) #2.3 | 3 months postoperatively
  The Expanded Prostate cancer Index Composite for Clinical Practice is a questionnaire to measure urinary, bowel,sexual and hormonal function of the patient's prostate cancer quality of life. The questionnaire is scored by the sum of the following scores: Urinary Incontinence symptom score, Urinary Irritation/Obstructive symptom score, Bowel Symptom score, Vitality/Hormonal symptom score and the overall prostate cancer quality of life score. The range of the score varies from 0 (best possible outcome) to 60 (worst possible outcome).
Expanded Prostate cancer Index Composite for Clinical Practice (EPIC-CP) #2.4 | 6 months postoperatively
  The Expanded Prostate cancer Index Composite for Clinical Practice is a questionnaire to measure urinary, bowel,sexual and hormonal function of the patient's prostate cancer quality of life. The questionnaire is scored by the sum of the following scores: Urinary Incontinence symptom score, Urinary Irritation/Obstructive symptom score, Bowel Symptom score, Vitality/Hormonal symptom score and the overall prostate cancer quality of life score. The range of the score varies from 0 (best possible outcome) to 60 (worst possible outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada